CLINICAL TRIAL: NCT02106325
Title: A Randomized, Double-Blinded Controlled Trial of an N-Methyl D-Aspartate Antagonist as a Rapidly-Acting Antidepressant in Depressed Emergency Department Patients
Brief Title: Ketamine as a Rapidly-Acting Antidepressant in Depressed Emergency Department Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-00794
Record Dates: First submitted 2013-12-12; First posted 2014-04-08 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Depression
Keywords: Ketamine; Ketlar; Depression; Antidepressants; Treatment; Acute
MeSH Terms: conditions — Depression | interventions — Ketamine; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): IV Ketamine .25mg/kg
  Interventions: Drug: Ketamine
- Diphenhydramine (Placebo Comparator): 25mg Diphenhydramine
  Interventions: Drug: Diphenhydramine

INTERVENTIONS:
Drug: Ketamine — IV of Ketamine (.25mg/kg)
  Other Names: Other names for ketamine: ketalar
  Arms: Ketamine
Drug: Diphenhydramine — Intravenous Diphenhydramine (25mg) at the time of presentation to Emergency Department
  Other Names: Other names for diphenhydramine: benadryl
  Arms: Diphenhydramine

SUMMARY:
Investigators will conduct a trial to evaluate the use of Ketamine as an alternate treatment for people with Major Depressive Disorder. This study plans to explore the potential that Ketamine's rapid antidepressant action holds for improving outcomes in patients presenting to the Emergency Department with severe depression. Since this is a controlled trial we will use an IV of Ketamine or and equivalent volume of Diphenhydramine. Subjects will be randomly assigned to receive Ketamine or Benadryl. Investigators will then compare measures of mood pre- and post-infusion in the Emergency Department. To supplement self-reported measures of depressive symptoms(e.g. mood), investigators will obtain objective measures of the biological aspects of Major Depressive Disorder.

DETAILED DESCRIPTION:
To explore the use of ketamine as a potential rapidly-acting antidepressant (RAA) for Emergency Department (ED) patients with major depressive disorder (MDD).

Investigators will conduct a randomized controlled study to evaluate the rapidity and persistence of antidepressant effects of a single sub-anesthetic dose of intravenous (IV) ketamine (0.25mg/kg) or an equivalent volume of diphenhydramine (25mg) delivered IV over 1-2 minutes, by comparing measures of mood pre- and post-infusion in Emergency Department (ED) patients with MDD. Subjects will be randomly assigned (1:1) to receive a bolus of ketamine or diphenhydramine. To supplement self-reported measures of depressive symptoms (e.g., mood, suicidal ideation, etc.), investigators will obtain objective measures of heart rate and heart rate variability, measure serum levels of the pro- and anti-inflammatory cytokines (interleukin IL-1, IL-2, IL-6, IL-8, IL-10, IL-12, and tissue necrosis factor, TNF-α), which have been shown to play an important role in stress, depression and suicidal behavior. In addition, investigators will obtain serum levels of brain derived neurotrophic factor (BDNF) because reduced serum BDNF has been described during acute depressive episodes in patients with MDD, with reports of rescue effects following treatment with various antidepressants and with ketamine (Aydemir 2005, Gervasoni 2005, Karege 2002, Karege 2005, Duncan 2013, Shimizu 2003). Investigators will also measure serum magnesium levels, as these have been shown to correlate in a predictive manner with response to conventional antidepressants (Camardese 2012), and there are data to suggest that ketamine's efficacy in treatment-resistant depression could be related to a relative magnesium deficiency in such patients (Murck 2013).

This study will allow investigators to determine to what extent low-dose ketamine, an N-Methyl-D-Aspartate (NMDA) antagonist, achieves a rapid reduction in symptoms for severely depressed ED patients with or without suicidal ideation. For decades, much higher doses of IV ketamine (1-2mg/kg) have been used routinely in the ED as a dissociative anesthetic (Green 2011). In 2011, an open-label study was the first published of the use of low dose ketamine (0.2mg/kg), administered by rapid intravenous infusion, in the ED setting for acutely depressed patients which demonstrated its feasibility, safety, preliminary efficacy and acceptability to both ED patients and staff (Larkin 2011). One long-term goal of this research is to expand treatment options available to depressed ED patients that mitigate the need for inpatient admission and serve as a safety bridge to future out-patient treatment for major depression. As an adjunct to standard treatment, low-dose NMDA receptor antagonists have the potential to positively impact: ED waiting times; repeat visits to the ED; short-term risk of suicide attempts; length of stay on inpatient units and the need for hospital admissions for many acutely depressed patients.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable as determined by the medical physician
* Meets criteria for Major Depressive Disorder (MDD) based on a structured clinical Interview (MINI International Neuropsychiatric Interview).
* Reports symptoms of severe depression at the time of presentation, defined as a score of 24 or greater on the MADRS.
* Patients for whom a psychiatric evaluation and disposition decision has been made by emergency psychiatry staff to admit to an inpatient psychiatric unit at Bellevue Hospital Center or NYU Tisch Hospital.
* Each subject must have a level of understanding sufficient to sign an informed consent stating that the treatment being offered is not FDA approved for the treatment of depression and is being provided as an off-label option.

Exclusion Criteria:

* Pregnancy
* Inability to read or understand English
* Current clinical signs of intoxication or delirium at time of study intervention
* Overdose, within previous 24 hours, of any agent which would impair ketamine metabolism
* Lifetime misuse/abuse of ketamine, phencyclidine (PCP),or related substances
* Lifetime history of psychotic spectrum illness
* First-degree relative with history of psychotic illness
* Lifetime diagnosis of borderline personality disorder, or as confirmed by assessment using items #90-104 of the SCID-II (for DSM-IV).
* Subjects with clinically significant abnormal findings as determined by medical history, physical examination, vital signs (blood pressure, heart rate, and respiration rate), O2 saturation measure, 12-lead ECG, clinical laboratory tests (CBC, chemistry panel, thyroid function tests), urine drug screen, and urine pregnancy test (for females of childbearing potential only).
* Clinically unstable medical, surgical or neurological conditions at ED presentation
* History of stroke or intracranial hypertension
* History of glaucoma
* Subjects with one or more seizures without a clear and resolved etiology
* Current NMDA antagonist medications (eg. Amantadine, Rimantadine, Lamotrigine, Memantine, Dextromethorphan)
* Known hypersensitivity to ketamine or amantadine
* Anti-psychotic medications (Typicals or Atypicals), with the exception of low-dose quetiapine (total daily dose of 100mg or less).
* Actively trying to commit suicide, even in a hospital setting
* Current homicide risk
* Unable or unwilling to give informed consent according to HIC guidelines
* Unable or unwilling to provide 2 contact phone numbers or be followed up per study protocol.
* Previous enrollment in this study.
* Concurrent enrollment in a research protocol investigating experimental pharmacologic treatments for depression at this or any other institution.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-12; Primary Completion 2016-02 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ross, MD, Principal Investigator — NYU Langone Health; K. Casey Paleos, MD, Study Chair — New York Unversity School of Medicine
Locations (2):
- United States (2):
  - Bellevue Hospital Center, New York, New York
  - NYU Langone Medical Center/Tisch Hospital, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Phase 1
Arm/Group | Ketamine | Diphenhydramine
Started | 5 | 3
Completed | 3 | 1
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2
Period: Phase 2
Arm/Group | Ketamine | Diphenhydramine
Started | 4 | 4
Completed | 2 | 1
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3
Period: Phase 3
Arm/Group | Ketamine | Diphenhydramine
Started | 2 | 3
Completed | 0 | 2
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Diphenhydramine | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Full Range); unit: years] | 40 [22 to 57] | 31 [22 to 48] | 38 [22 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Effects of Ketamine on Depressive Symptomatology by Measuring Change in Score on the Montgomery-Asberg Depressive Rating Scale
Description: 40 Minutes Post Infusion, The MADRS-S instrument has nine questions, with an overall score ranging from 0 to 54 points.
  0 to 6 - normal /symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ketamine | Diphenhydramine
Number analyzed (Participants) | 11 | 10
units on a scale | 28.82 (2.95) | 25.20 (3.10)

2. Primary Outcome: Beck Depression Inventory-II (BDI-II)
Description: BDI-II items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63.
  0-13 Indicates minimal depression 14-19 Indicates mild depression 20-28 Indicates Moderate depression 29-63 Indicates Severe depression
Time Frame: 120 min post-infusion
Measure: Mean (Standard Error); unit: Scored units on a scale
Arm/Group | Ketamine | Diphenhydramine
Number analyzed (Participants) | 11 | 10
Scored units on a scale | 20.00 (3.94) | 24.72 (4.06)

3. Primary Outcome: Hamilton Depression Scale (Ham-D)
Description: Although the HAM-D form lists 21 items, the scoring is based on the first 17. It generally takes 15-20 minutes to complete the interview and score the results. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2.
  Sum the scores from the first 17 items 0-7= Normal 8-13= Mild Depression 14-18= Moderate Depression 19-22= Severe Depression >23= Very Severe Depression
Time Frame: 4-6 hours post-infusion
Measure: Mean (Standard Error); unit: Scored units on a scale
Arm/Group | Ketamine | Diphenhydramine
Number analyzed (Participants) | 11 | 10
Scored units on a scale | 21.48 (2.08) | 17.00 (2.26)

4. Secondary Outcome: Change in Treatment Alliance Score
Description: The I-TAS is a 10-item, Likert-style rating scale designed to assess a patient's composite treatment alliance as it develops across multi-disciplinary treatment components. The I-TAS was intended to measure the primary alliance factors identified by Hatcher and Barends (1996) of bond, goals and collaboration. Each question is scored on a scale of 0 (Completely False) to 6 (Completely True). Total scores on the ITAS range from 0 to 60, with higher scores representing greater alliance with the treatment team (better outcome). The reported score is an average of each participant's total score on the ITAS.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Error); unit: Scored units on a scale
Arm/Group | Ketamine | Diphenhydramine
Number analyzed (Participants) | 11 | 10
Scored units on a scale | 43.52 (3.69) | 53.15 (4.17)

5. Secondary Outcome: Beck Scale for Suicidal Ideation (BSSI)
Description: as for outcome 2
Time Frame: 40 minutes post-infusion
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ketamine | Diphenhydramine
Number analyzed (Participants) | 11 | 10
units on a scale | 1.58 (1.40) | 1.08 (1.42)

6. Secondary Outcome: Montgomery-Åsberg Depression Rating Scale Suicide Ideation Item (MADRS-SI)
Description: as for outcome 1
Time Frame: 40 minutes post-infusion
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ketamine | Diphenhydramine
Number analyzed (Participants) | 11 | 10
units on a scale | 0.83 (0.46) | 0.75 (0.40)

7. Secondary Outcome: Length of Inpatient Stay
Time Frame: 2 Weeks Post-infusion
Measure: Mean (Standard Error); unit: Days
Arm/Group | Ketamine | Diphenhydramine
Number analyzed (Participants) | 11 | 10
Days | 6.33 (1.32) | 7.80 (1.25)

8. Secondary Outcome: Outpatient Follow-up Compliance
Description: Scoring System: 0= not compliant, 1=compliant
Time Frame: 1 Day
Measure: Mean (Standard Error); unit: units on follow up compliance scale
Arm/Group | Ketamine | Diphenhydramine
Number analyzed (Participants) | 11 | 10
units on follow up compliance scale | 0.73 (.14) | .70 (.14)

9. Secondary Outcome: Inpatient Treatment Alliance Scale (ITAS)
Description: as for outcome 4
Time Frame: 7 days post-infusion
Measure: Mean (Standard Error); unit: Scored units on ITAS Scale
Arm/Group | Ketamine | Diphenhydramine
Number analyzed (Participants) | 11 | 10
Scored units on ITAS Scale | 43.52 (3.69) | 53.15 (4.17)

ADVERSE EVENTS:
Arm/Group | Ketamine | Diphenhydramine
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/10
Other Adverse Events (participants affected / at risk) | 8/11 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=11) | Diphenhydramine (N=10)
Psychosis and Suicidality (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=11) | Diphenhydramine (N=10)
Tiredness (General disorders) | 1 (1) | 3 (3)
Perceptual Disturbance (General disorders) | 2 (2) | 2 (2)
Headache (General disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 2 (2) | 1 (1)
Toe Numbness (General disorders) | 0 (0) | 1 (1)
GI Distress (General disorders) | 2 (2) | 0 (0)
Elevated Systolic BP (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes